CLINICAL TRIAL: NCT06059807
Title: A Cone-Beam Computed Tomography Evaluation of Root Resorption After Maxillary Expansion Using Hyrax and Hybrid Hyrax Appliances (Expanders)
Brief Title: Root Resorption After Maxillary Expansion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Mohamed Taher Mohamed Abo Ghalia, Principle investigator, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: expanders
Record Dates: First submitted 2023-09-14; First posted 2023-09-29 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Maxillary Expansion
Keywords: expanders
MeSH Terms: interventions — Palatal Expansion Technique

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hyrax group (Experimental)
  Interventions: Device: maxillary expansion
- hybrid hyrax group (Experimental)
  Interventions: Device: maxillary expansion

INTERVENTIONS:
Device: maxillary expansion — Maxillary Expansion Using Hyrax and Hybrid Hyrax Appliances

SUMMARY:
The aim of this study will to evaluate the root resorption after RME by hyrax and hybrid hyrax appliances by using of cone beam computed tomography .

ELIGIBILITY:
Inclusion Criteria:

1. skeletal maxillary transvers deficiency
2. unilateral or bilateral posterior crossbite
3. negative buccal corridor
4. patient with good oral hygiene
5. patient with no previous orthodontic treatment
6. no systemic disease

Exclusion Criteria:

1. craniofacial congenital anomalies
2. a history of periodontal disease
3. incomplete treatment records

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Change in root resorption after maxillary expansion | 12 weeks following end of treatment
  A Cone-Beam Computed Tomography Evaluation of Root Resorption After Maxillary Expansion Using Hyrax and Hybrid Hyrax Appliances

REFERENCES:
- [Result] Miranda F, Cunha Bastos JCD, Magno Dos Santos A, Janson G, Pereira Lauris JR, Garib D. Dentoskeletal comparison of miniscrew-anchored maxillary protraction with hybrid and conventional hyrax expanders: A randomized clinical trial. Am J Orthod Dentofacial Orthop. 2021 Dec;160(6):774-783. doi: 10.1016/j.ajodo.2021.02.017. Epub 2021 Sep 9. PMID 34509329
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/34509329/